CLINICAL TRIAL: NCT01400022
Title: A Randomized Clinical Study Comparing Topical 0.05% Clobetasol Propianate in Vaseline With UVA-1 Phototherapy in the Treatment of Vulvar Lichen Sclerosus
Brief Title: Topical 0.05% Clobetasol Propionate in Vaseline Versus UVA-1 Phototherapy in Vulvar Lichen Sclerosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, AKreuter, Prof. Dr., Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RUB-125
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: lichen; sclerosus; genital; vulvar; UVA1
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Cortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cortisone (Active Comparator)
  Interventions: Other: Cortisone
- UVA1 phototherapy (Experimental)
  Interventions: Other: UVA1 phototherapy

INTERVENTIONS:
Other: UVA1 phototherapy — The UVA1-phototherapy is conducted 4 times per week over a period of 3 months. A UVA1-irradiation device of the company Sellamed, Gevelsberg (Germany) is used. The radiation intensity is 24 mW/cm ². The distance between radiation source and irradiation area is approximately 25 cm. Over five sessions, the UVA1 dose is increased slowly, starting with 10 J/cm ² in the first, 20 J/cm ² in the second and 30 J/cm ² in the third, 40 J/cm ² in the fourth, and from the fifth session 50 J/cm ². Additionally, a topical treatment with vaseline album once daily can be applied after irradiation (not before irradiation).
  Arms: UVA1 phototherapy
Other: Cortisone — Clobetasol propionate (0.05%) in white vaseline is applied thinly once daily. The duration of treatment is 3 months.
  Arms: Cortisone

SUMMARY:
Lichen sclerosus is a rare, chronic cutaneous disorder with a predilection for the genital area. Any age group may be affected, although it is seen more often in postmenopausal women. The current gold standard treatment is topical ultrapotent corticosteroids such as clobetasol.

Here we compare UVA1 phototherapy with 0,05% clobetasol propionate in vaseline for the treatment of vulvar lichen sclerosus.

DETAILED DESCRIPTION:
Genital lichen sclerosus is a rare chronic inflammatory connective tissue disease. The association with other autoimmune diseases and the detection of autoantibodies against ECM-1 point to an autoimmune genesis. Genital lichen sclerosus typically affects women around and after the menopause. Common sites of affection are the vulva (clitoris and labia majora) and the anus in women, the prepuce and the glans penis in men. Skin lesions include ivory-white, atrophic, porcelain-like plaques with a tendency to atrophy and fissures in the advanced stages.

First-line therapy for genital lichen sclerosus in the active, inflammatory phase is the use of topical glucocorticoids. Alternatively, topically applied hormone-containing emollients and topical calcineurin inhibitors are widely used. However, the use of topical corticosteroids is because of the associated long-term side effects (atrophy, striae) limited.

In the treatment of localized scleroderma (morphea), a similar sclerosing disease, the use of ultraviolet radiation (UVA1) has proved highly effective. After a pilot study, the high-dose UVA1 phototherapy (120 J / cm ²) was significantly more effective was a low-dose UVA1 (20 J / cm ²), however no difference could be found in subsequent studies. Meanwhile, the medium-dose UVA1 phototherapy in circumscribed scleroderma has been determined as the most effective therapy regime and is included in the german dermatological guidelines (see also AWMF guideline for diagnosis and therapy of circumscribed scleroderma at: http://www.uni-duesseldorf.de/awmf/ll/013- 066.htm).

ELIGIBILITY:
Inclusion Criteria:

* patients with genital lichen sclerosus
* Age > 18 years
* Willingness to participate in this study
* No topical steroids within the last 4 weeks

Exclusion Criteria:

* Age < 18 years
* Known photodermatosis (eg, solar urticaria, polymorphous light eruption)
* Known genodermatosis with UV-sensitivity
* Treatment with photosensitizing drugs
* History of skin cancer
* significant UV exposure 3 months before study entry
* application of UV radiation therapies outside of the study conducted by UV irradiation: as: PUVA, UVA (including UVA1), UVB (including SEA) in the last 4 weeks before study entry or during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Clinical improvement during UVA1/cortisone treatment | 6 months follow-up
  Clinical improvement during UVA1/cortisone treatment using an investigator score measuring hypopigmentation, sclerosis, atrophy, hyperkeratosis, erosions, edema, erythema in a numerical scale as to be rated followed: 0 = absent, 1 = mild, 2 = moderate, 3 = severe. The total score is then calculated respectively from the sum of individual scores (max. 21 points).

SECONDARY OUTCOMES:
subjective patient score | until 6 months follow-up
  a subjective patient-score to measure burning, pain and itch using a visual analogue scale with score from 0 (absent) to 10 (most severe imaginable)
Influence on Quality of Life | until 6 months follow-up
  Measuring the influence of the disease on the Quality of Life using a qualified Questionnaire on Quality of Life in Dermatology: Skindex-29
Colorimetry | baseline and after 3 months of treatment
  Objective measurement of colour to determine erythema, severity of white patches.
Ultrasound to determine the severity of the sclerosis | baseline and after 3 months of treatment
  A 22MHz Ultrasound of the involved area is performed at the baseline and after 3 months of therapy to determine the severity of the sclerosis
Immunological, RT-PCR and histological parameters in skin biopsies | baseline and after 3 months of treatment
  Measuring several immunohistochemical, RT-PCR and serological parameters in skin and blood, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kreuter, MD, Prof., Principal Investigator — Ruhr University Bochum; Sarah Terras, MD, Principal Investigator — Ruhr University Bochum; Thilo Gambichler, MD, Principal Investigator — Ruhr University Bochum
Locations (1):
- Department of Dermatology, Ruhr University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Terras S, Gambichler T, Moritz RK, Stucker M, Kreuter A. UV-A1 phototherapy vs clobetasol propionate, 0.05%, in the treatment of vulvar lichen sclerosus: a randomized clinical trial. JAMA Dermatol. 2014 Jun;150(6):621-7. doi: 10.1001/jamadermatol.2013.7733. PMID 24696010